CLINICAL TRIAL: NCT00402285
Title: The Molecular Effects of Nutrition Supplements (MENS) Prostate Study
Brief Title: Lycopene or Omega-3 Fatty Acid Nutritional Supplements in Treating Patients With Stage I or Stage II Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CDR0000505501; UCSF-03553; UCSF-H5664-22834-04A
Record Dates: First submitted 2006-11-20; First posted 2006-11-22 (Estimated); Results first posted 2013-05-16 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- lycopene supplement (Active Comparator): Two 15mg lycopene capsules daily for 3 months.
  Interventions: Dietary Supplement: lycopene supplement
- fish oil supplement (Active Comparator): 1g fish oil capsule daily for 3 months.
  Interventions: Dietary Supplement: fish oil supplement
- placebo (Placebo Comparator): placebos for lycopene and fish oil.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: lycopene supplement
  Arms: lycopene supplement
Dietary Supplement: fish oil supplement
  Arms: fish oil supplement
Other: Placebo — placebos for lycopene and fish oil.
  Arms: placebo

SUMMARY:
RATIONALE: The use of lycopene, a substance found in tomatoes, or omega-3 fatty acid nutritional supplements may keep cancer from growing in patients with prostate cancer.

PURPOSE: This randomized clinical trial is studying lycopene to see how well it works compared to omega-3 fatty acids or a placebo in treating patients with stage I or stage II prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare gene expression in normal prostate tissue (at baseline and after treatment) of patients with stage I or II adenocarcinoma of the prostate treated with lycopene vs omega-3 fatty acid nutritional supplements vs placebo.

Secondary

* Determine new candidate molecular targets for lycopene and omega-3 response pathways.
* Correlate baseline gene expression patterns, determined by cDNA array analysis, with self-reported dietary intake.
* Correlate gene expression patterns with progression or lack of progression at 12 months after study entry.
* Determine if lycopene or omega-3 supplements affect the incidence of tumor progression.

OUTLINE: This is a randomized, placebo-controlled study. Patients are stratified according to dietary intake of tomato and fish (low tomato [< 4 servings/week], low fish [< 2 servings/week] vs low tomato, high fish [≥ 2 servings/week] vs high tomato [≥ 4 servings/week], low fish vs high tomato, high fish). Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients maintain normal diet and receive oral omega-3 fatty acids placebo 3 times daily and lycopene placebo twice daily.
* Arm II: Patients receive oral lycopene twice daily and oral omega-3 fatty acids placebo 3 times daily.
* Arm III: Patients receive oral lycopene placebo twice daily and oral omega-3 fatty acids 3 times daily.

In all arms, treatment continues for up to 90 days or until post-treatment biopsy is scheduled (a maximum of 104 days) in the absence of disease progression.

Patients complete a dietary questionnaire at baseline and then for 3 days each month during study therapy. Quality of life is assessed at baseline and at 3 months.

Prostate tissue needle biopsies and blood samples are collected at baseline and at 3 months. Tissue and blood samples are examined for lycopene and omega-3 fatty acids (treatment compliance), omega-6 fatty acids, insulin-like growth factor (IGF)-1, IGF binding protein-5, and cyclooxygenase-2 gene by polymerase chain reaction, cDNA microarray hybridization, and other gene expression assays.

After completion of study treatment, patients are followed every 3 months for 2 years.

PROJECTED ACCRUAL: A total of 114 patients will be enrolled in this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate meeting the following criteria:

  * Newly diagnosed disease
  * Small cell acinar type
  * Gleason score ≤ 6 with no pattern 4 or 5 histology

    * Gleason pattern 4 seen as a microfocus (< 2 mm in length) allowed
  * Stage I-II (T1 or T2a) disease
* Must have had an extended pattern biopsy (defined as 8+ cores) within the past 2 years

  * Patients meeting all of the eligibility criteria except for the aforementioned extended pattern biopsy within the past two years may enroll in the study if they have an extended pattern clinical biopsy scheduled no more than 6 weeks before beginning study treatment AND are willing to have an additional 4 biopsy cores
* No more than 33% of biopsy cores positive

  * 33% or more of biopsy cores positive due to microfoci of adenocarcinoma allowed
* No more than 50% of the length of a tumor core involved by carcinoma
* Watchful waiting planned as primary treatment strategy
* Must have 3 serum prostate-specific antigen (PSA) level readings taken ≥ 2 weeks apart over the past year

  * PSA ≤ 10.0 ng/mL

    * PSA < 15 ng/mL in patients with benign prostatic hyperplasia or prostatitis allowed
  * PSA doubling time ≥ 3 months

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 3 months
* ECOG performance status 0-2
* No history of allergic reactions attributed to tomatoes, fish, soybean oil, gelatin capsules, or compounds of similar chemical or biologic composition to lycopene (carotenoids) or fish oil (omega-3 fatty acids)
* No uncontrolled intercurrent illness including, but not limited to, the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situations that would limit study compliance

PRIOR CONCURRENT THERAPY:

* No prior or concurrent treatment for prostate cancer, including surgery, radiation, hormonal therapy (e.g., leuprolide acetate, bicalutamide, flutamide, goserelin, megestrol, nilutamide, diethylstilbestrol/estrogen), chemotherapy, PC-SPES, or investigational agents
* More than 4 weeks since prior and no concurrent lycopene, fish oil (omega-3 fatty acids), or any other preparation intended to supplement levels of omega-3 unsaturated fatty acids
* More than 4 weeks since prior and no concurrent finasteride, dutasteride, saw palmetto or any other herbal/nutritional preparation indicated to affect hormone levels
* More than 1 month since prior nonsteroidal anti-inflammatory drugs (NSAIDs), cyclooxygenase-2 (COX-2) inhibitors, and/or aspirin for > 7 days duration
* No concurrent NSAIDs, COX-2 inhibitors, or aspirin

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2003-04; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter R. Carroll, MD, Study Chair — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States

REFERENCES:
- [Result] Magbanua MJ, Roy R, Sosa EV, Weinberg V, Federman S, Mattie MD, Hughes-Fulford M, Simko J, Shinohara K, Haqq CM, Carroll PR, Chan JM. Gene expression and biological pathways in tissue of men with prostate cancer in a randomized clinical trial of lycopene and fish oil supplementation. PLoS One. 2011;6(9):e24004. doi: 10.1371/journal.pone.0024004. Epub 2011 Sep 1. PMID 21912659
- [Derived] Magbanua MJ, Richman EL, Sosa EV, Jones LW, Simko J, Shinohara K, Haqq CM, Carroll PR, Chan JM. Physical activity and prostate gene expression in men with low-risk prostate cancer. Cancer Causes Control. 2014 Apr;25(4):515-23. doi: 10.1007/s10552-014-0354-x. Epub 2014 Feb 7. PMID 24504435

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potentially eligible men identified at Urologic Oncology clinic at Helen Diller Family Comprehensive Cancer Center San Francisco starting in 2003.
Groups:
- Lycopene Supplement: two 15mg lycopene soft gel capsules daily (Lyc-O-Mato). men took lycopene & placebo for fish oil.
- Fish Oil Supplement: three 1g fish oil capsules daily including 1,098mg EPA & 549mg DHA fatty acid (Roche).
  men took fish oil & placebo for lycopene.
- Placebo: men took placebo for lycopene & placebo for fish oil.
Period: Overall Study
Arm/Group | Lycopene Supplement | Fish Oil Supplement | Placebo
Started | 29 | 27 | 28
Completed | 22 | 21 | 26
Not Completed | 7 | 6 | 2
Not completed — insufficient RNA quality | 7 | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lycopene Supplement | Fish Oil Supplement | Placebo | Total
Number analyzed (Participants) | 29 | 27 | 28 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (7) | 62 (8) | 59 (8) | 61 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 29 | 27 | 28 | 84

OUTCOME MEASURES:

1. Primary Outcome: Changes in Normal Prostate Tissue Gene Expression Between the Baseline and 3-month Biopsies in IGF -1 and COX -2
Description: Comparisons of the change in deltaCT were between the placebo and Lycopene arms for IGF-1 and IGF-1R and between the placebo and fish oil arms for COX-2. Data in the table are mean changes in qRTPCR gene expression (normalized to GUSb) for IGF1, Cox2, and IGF1R.
Time Frame: baseline through 3 month
Population: 1 ppt randomized to fish oil had un-evaluable COX-2 at 3 months.
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | Lycopene Supplement | Fish Oil Supplement | Placebo
Number analyzed (Participants) | 22 | 20 | 26
fold change
  IGF-1 | 0.05 (1.32) | NA (NA) — we did not measure IGF for fish oil | 0.02 (1.22)
  COX-2 | NA (NA) — we did not measure COX-2 for lycopene | 0.39 (1.98) | 0.40 (2.19)
  IGF-1R | 0.20 (3.00) | NA (NA) — we did not measure IGF for fish oil | 0.74 (2.86)

ADVERSE EVENTS:
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/84
Other Adverse Events (participants affected / at risk) | 0/84

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No